CLINICAL TRIAL: NCT02922569
Title: Home-Based, Online, Mindfulness and Cognitive Training for Soldiers and Veterans With TBI
Acronym: CogMind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-0616-16; AZ150059 (Other: eBRAP Log Number)
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training and mindfulness training requiring a total maximum of 60 treatment sessions, up to 5 sessions per week, 40 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training; Other: Mindfulness Training
- Active Comparator (Active Comparator): Commercially available computerized training and traumatic brain injury information session requiring a total maximum of 60 treatment sessions, up to 5 sessions per week, 40 minutes per session.
  Interventions: Other: Commercially available computerized training; Other: Traumatic Brain Injury Information Session

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Thirty minutes of training on computerized exercises that targets processing speed, memory and attention.
  Arms: Experimental Treatment
Other: Commercially available computerized training — Thirty minutes of training on computerized, casual video games.
  Arms: Active Comparator
Other: Mindfulness Training — Ten minutes of using an online training course that teaches skills to help overcome ongoing life stressors.
  Arms: Experimental Treatment
Other: Traumatic Brain Injury Information Session — Ten minutes of viewing traumatic brain injury related news, information, and programs.
  Arms: Active Comparator

SUMMARY:
This study is a parallel arm, double-blind, randomized, controlled clinical trial to assess the safety and efficacy of an experimental software program designed to improve cognitive functions versus a computer-based software control. Both the study and the software being investigated meet the criteria of Non-Significant Risk.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effects of combination of mindfulness training (MT) and adaptive cognitive training (CT) on the cognitive abilities, functional status and quality of life of soldiers and veterans diagnosed with traumatic brain injury (TBI, also referred to as a concussion, or blast exposure), as compared to a computer-based control.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants must have diagnosis of mild traumatic brain injury (mTBI) confirmed by Ohio State University TBI Identification Method-Short Form (OSU TBI-ID-SF)
* Participants must have persistent cognitive dysfunction confirmed by an objective measure (Automated Neuropsychological Assessment Metrics (ANAM) TBI Battery with a score at least one standard deviation below the age-adjusted norm for a military sample) or a subjective measure (Ruff Neurobehavioral Inventory (RNBI) with a score of greater than 70 on any of the four cognitive scales (Attention, Memory, Language, Executive)
* Participants must be at least six months out from their most recent traumatic brain injury (TBI), concussion, and/or blast exposure
* Participant must be a fluent English speaker
* Participants must score ≥ 70 on the Wechsler Test of Adult Reading (WTAR)
* Participants must have adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a computer mouse

Exclusion Criteria:

* Participants with history of TBI with loss of consciousness for more than 24 hours or post-traumatic amnesia for more than 7 days
* Participants with a history of penetrating head wounds
* Participants who are in-patients
* Participants with a diagnosis of an illness or condition with known cognitive consequences (e.g., schizophrenia, bipolar disorder, cancer, multiple sclerosis)
* Participants with active suicidal ideation with specific plan and intent or suicide-related behaviors within 2 months of consent as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Participants showing signs of intoxication due to current substance abuse (including alcohol and/or illegal drugs) during any in person visit
* Participants with clinically significant visual field deficits
* Participants judged to be lacking effort
* Participants with problems performing assessments or comprehending or following spoken instructions
* Participants enrolled in a concurrent clinical trial involving an investigational pharmaceutical, nutraceutical, medical device, or behavioral treatment for TBI that could affect the outcome of this study
* Participant with self-reported claustrophobia or physician-reported implanted devices (e.g. pacemakers, cochlear implants, aneurysm clips, etc.) and pregnant women will not be able to participate in MRI portion of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Changes in performance on global cognitive composite score | At 3 months and at 6 months
  Change in performance on global cognitive composite score based on the average of all normalized assessment measures.

SECONDARY OUTCOMES:
Changes in performance on processing speed composite score | At 3 months and at 6 months
  Change in performance on processing speed will be measured using the composite score created by averaging the z-scores of Pattern Comparison, Letter Comparison, and Digit Symbol Coding tasks.
Changes in performance on memory composite score | At 3 months and at 6 months
  Change in performance on memory will be measured using the composite score created by averaging the z-scores of N-Back task, Spatial Working Memory task, WAIS-IV Digit Span and Rey Auditory Verbal Learning Test (RAVLT).
Changes in performance on executive function composite score | At 3 months and at 6 months
  Change in performance on executive function will be measured using the composite score created by averaging the z-scores for the Trail Making, Flanker, and Stroop tasks.
Change in functional performance | At 3 months and at 6 months
  Between-group magnitude of change in sum time of all tasks in the Timed Instrumental Activities of Daily Living (TIADL). Higher scores indicate greater impairment in functional performance.
Change in TBI functional status | At 3 months and at 6 months
  Between-group magnitude of change in overall T-score using the self-report measure, Mayo-Portland Adaptability Inventory (MPAI-4). The overall T-score range is -38 to 106. Higher scores indicate more severe TBI functional status.
Changes in brain function | At 3 months
  Change in resting state functional connectivity will be measured by 12-minutes of resting state functional MRI. Participants will be instructed to keep their eyes open and maintain attention on a white fixation cross on a black screen.
Changes in brain structure | At 3 months
  Structural brain integrity will be measured with a high resolution 3D T1-weighted scan with good gray/white matter contrast and a complementary high-resolution T2-weighted anatomical scan.
Changes in task-related brain activation | At 3 months
  Change in functional connectivity and brain activation will be measured while performing N-Back Task.

OTHER OUTCOMES:
Change in Neurobehavioral Symptoms | At 3 months and at 6 months
  Between-group magnitude of change in sum score using the self-report measure, Neurobehavioral Symptoms Index (NSI). The scoring range is 0-88. Higher scores indicate more severe neurobehavioral symptoms.
Change in PTSD Symptoms | At 3 months and at 6 months
  Between-group magnitude of change in sum score using the self-report measure, PTSD Checklist (PCL-5). The scoring range is 0-80. Higher scores indicate more severe PTSD symptoms
Change in Depressive Symptoms | At 3 months and at 6 months
  Between-group magnitude of change in sum score using the self-report measure, Beck Depression Inventory (BDI-II). The scoring range is 0-63. Higher scores indicate more severe depressive symptoms.
Change in Health-Related Quality of Life | At 3 months and at 6 months
  Between-group magnitude of change in sum score using the self-report measure, Quality of Life after Brain Injury (QOLIBRI). The scoring range is 0-100. Lower scores indicate lower quality of life.
Change in Executive Function Symptoms | At 3 months and at 6 months
  Between-group magnitude of change in After total T-score using the self-report measure, Frontal Systems Behavior Scale (FrSBe). Raw scores are converted to age- and education-corrected T-scores. The mean T-score is 50, scores greater than 65 are considered clinically significant.
Change in Cognitive Symptoms | At 3 months and at 6 months
  Between-group magnitude of change in sum score using the self-report measure, Cognitive Failures Questionnaire (CFQ). The scoring range is 0-100. Higher scores indicate more severe cognitive symptoms.
Change in Work/School Status | At 3 months and at 6 months
  Change in total score using the self-report questionnaire about their work/school status.
Change in Physical Activity | At 3 months
  Change in total score based on weekly self-report dairy about physical activity during training period.
Change in Diet | At 3 months
  Change in total score based on weekly self-report dairy about diet during training period.
Change in Social Activity | At 3 months
  Change in total score based on weekly self-report dairy about social activity during training period.
Change in Sleep | At 3 months
  Change in total score based on weekly self-report dairy about sleep during training period.
Change in Functional Abilities | At 3 months
  Change in total score based on weekly self-report dairy about functional abilities during training period.

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Lee, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Veterans Affairs Connecticut Health Care System, West Haven, Connecticut, United States